CLINICAL TRIAL: NCT01381900
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, 18-Week Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Alone or in Combination With a Sulphonylurea
Brief Title: A Efficacy, Safety, and Tolerability Study of Canagliflozin in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Alone or in Combination With a Sulphonylurea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018541; 28431754DIA3014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100mg (Experimental): Each participant will receive 100 mg of canagliflozin once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
  Interventions: Drug: Canagliflozin 100mg; Drug: Metformin; Drug: Sulphonylurea
- Canagliflozin 300mg (Experimental): Each participant will receive 300 mg of canagliflozin once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
  Interventions: Drug: Canagliflozin 300mg; Drug: Metformin; Drug: Sulphonylurea
- Placebo (Placebo Comparator): Each participant will receive matching placebo once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Sulphonylurea

INTERVENTIONS:
Drug: Placebo — Form=capsule, route=oral administration. One capsule once daily for up to 18 weeks after completing a single-blind placebo run-in period (1 placebo capsule once daily for up to 2 weeks).
  Arms: Placebo
Drug: Canagliflozin 100mg — Type=1, unit=mg, number=100, form=capsule, route=oral use. One capsule once daily for up to 18 weeks after completing a single-blind placebo run-in period (1 placebo capsule once daily for up to 2 weeks).
  Arms: Canagliflozin 100mg
Drug: Canagliflozin 300mg — Type=1, unit=mg, number=300, form=capsule, route=oral use. One capsule once daily for up to 18 weeks after completing a single-blind placebo run-in period (1 placebo capsule once daily for up to 2 weeks).
  Arms: Canagliflozin 300mg
Drug: Metformin — The participant's stable dose of background therapy of metformin should be continued throughout the study.
Drug: Sulphonylurea — The participant's stable dose of background therapy of metformin plus sulphonylurea should be continued throughout the study.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of the addition of canagliflozin relative to the addition of placebo in patients with inadequate glycemic control on metformin alone or in combination with a sulphonylurea.

DETAILED DESCRIPTION:
This is a double-blind (neither study staff or the patient will know the identity of the treatment assigned) study of canagliflozin where Chinese and other Asian adult patients with Type 2 Diabetes Mellitus (T2DM) who have inadequate glycemic control on metformin alone or in combination with a sulphonylurea (SU) will be randomized (assigned to 1 of 3 treatments by chance) to receive the addition of treatment with canagliflozin 100 mg once daily, canagliflozin 300 mg once daily, or matching placebo capsules (placebo is a treatment identical in appearance to canagliflozin but does not contain active drug). All patients will take orally (by mouth) 1 single-blind placebo capsule once daily before the first meal of the day for up to 2 weeks (last dose of single-blind placebo to be taken the day before the baseline (Day 1) visit. On Day 1, patients will take orally, once daily 1 capsule of canagliflozin 100 mg, canagliflozin 300 mg, or placebo before the first meal of the day for up to 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM with inadequate glycemic control on metformin monotherapy or on metformin in combination with an SU at protocol-specified doses and having HbA1c >=7.0% and <=10.5% at Week -2 are eligible for enrollment in the study.

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Has repeated (ie, 2 or more over a 1-week period) fasting plasma glucose (FPG) and/or fasting self-monitored blood glucose (SMBG) measurements >=270 mg/dL (15 mmol/L) during the pre-treatment phase, despite reinforcement of diet and exercise counseling
* History of a severe hypoglycemic episode within 6 months before screening
* History of or current illness considered to be clinically significant by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (25):
- China (20):
  - Baotou
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Harbin
  - Nanchang
  - Nanjing
  - Nanning
  - Shanghai
  - Shenyang
  - Shiyan
  - Siping
  - Suzhou
  - Tianjin
  - Wuxi
  - Xi'an
- Malaysia (3):
  - Kota Bharu
  - Kuala Selangor
  - Pulau Pinang
- Vietnam (2):
  - Hanoi
  - Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in Asian participants with type 2 diabetes mellitus who had inadequate glycemic control on a maximally effective or tolerated dose of metformin alone or metformin plus sulphonylurea (SU). It was conducted between 30 June 2011 and 21 December 2012 and recruited patients from 36 sites.
Pre-assignment Details: The study had two background treatment strata: 331 participants in the metformin alone stratum and 347 in the metformin plus SU. In total, 678 participants were randomly allocated to the 3 treatment arms, 676 received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set and the safety analysis set.
Groups:
- Placebo: Each participant received matching placebo once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
- Canagliflozin 100 mg: Each participant received 100 mg of canagliflozin once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
- Canagliflozin 300 mg: Each participant received 300 mg of canagliflozin once daily for 18 weeks with protocol-specified doses of metformin alone or metformin plus sulphonylurea.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 226 | 223 | 227
Completed | 217 | 214 | 215
Not Completed | 9 | 9 | 12
Not completed — Subject meets glycemic withdrawal crit. | 2 | 0 | 0
Not completed — Adverse Event | 4 | 6 | 7
Not completed — Noncompliance with study drug | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Early withdraw | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 226 | 223 | 227 | 676
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 184 | 187 | 186 | 557
  >=65 years | 42 | 36 | 41 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.35) | 56.5 (8.25) | 56.4 (9.21) | 56.3 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 99 | 114 | 314
  Male | 125 | 124 | 113 | 362
Region Enroll [Number; unit: participants]
  China | 213 | 210 | 213 | 636
  Malaysia | 3 | 5 | 4 | 12
  Vietnam | 10 | 8 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean change in HbA1c from baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 18
Population: Analysis used overall mITT analysis set (all randomized patients who received at least 1 dose of double-blind study drug). Last-observation-carried-forward method used for missing Week 18 values. Table includes only participants with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 226 | 223 | 227
Percent | -0.47 (0.096) | -0.97 (0.095) | -1.06 (0.095)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.51, 95% CI 2-sided [-0.644 to -0.367], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.59, 95% CI 2-sided [-0.731 to -0.453], Standard Error of Mean 0.071

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 18
Population: Analysis used overall mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 18 values. Table includes only participants with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 226 | 223 | 227
mg/dL | -0.40 (0.237) | -1.44 (0.236) | -1.83 (0.235)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.03, 95% CI 2-sided [-1.375 to -0.694], Standard Error of Mean 0.173
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -1.43, 95% CI 2-sided [-1.769 to -1.089], Standard Error of Mean 0.173

3. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 18
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 18 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Pecent change
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 226 | 223 | 227
Pecent change | -0.8 (0.4) | -2.9 (0.4) | -3.1 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.2, 95% CI 2-sided [-2.7 to -1.6], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.3, 95% CI 2-sided [-2.9 to -1.8], Standard Error of Mean 0.3

4. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) <7% at Week 18
Description: The table below shows the percentage of patients with HbA1c <7% at Week 18 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Day 1 (Baseline) and Week 18
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 226 | 223 | 227
Percentage of patients | 27.8 | 49.1 | 52.9
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 3.26, 95% CI 2-sided [2.09 to 5.09]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 3.99, 95% CI 2-sided [2.55 to 6.27]

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) <6.5% at Week 18
Description: The table below shows the percentage of patients with HbA1c <6.5% at Week 18 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Day 1 (Baseline) and Week 18
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 226 | 223 | 227
Percentage of patients | 11.7 | 21.6 | 25.3
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.45 to 4.48]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.88 to 5.75]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study, consisting of an 18-week double-blind treatment phase and a 4-week follow-up period.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any of the treatment arms during the study.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Serious Adverse Events (participants affected / at risk) | 4/226 | 5/223 | 4/227
Other Adverse Events (participants affected / at risk) | 22/226 | 27/223 | 27/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=226) | Canagliflozin 100 mg (N=223) | Canagliflozin 300 mg (N=227)
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=226) | Canagliflozin 100 mg (N=223) | Canagliflozin 300 mg (N=227)
Upper respiratory tract infection (Infections and infestations) | 14 | 7 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 20 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days